CLINICAL TRIAL: NCT03493685
Title: A Randomized, Multicenter, Double-blind, Parallel, Active-control Study of the Effects of Sparsentan, a Dual Endothelin Receptor and Angiotensin Receptor Blocker, on Renal Outcomes in Patients With Primary FSGS
Brief Title: Study of Sparsentan in Patients With Primary Focal Segmental Glomerulosclerosis (FSGS)
Acronym: DUPLEX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 021FSGS16010
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — sparsentan; Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- sparsentan for double-blind and open-label extension (Experimental): Sparsentan will be administered as a single oral dose; an initial dose of 400 mg daily titrating up to a target dose of 800 mg, daily
  Interventions: Drug: sparsentan
- Irbesartan (Active Comparator): Irbesartan will be administered as a single oral dose; an initial dose of 150 mg daily titrating up to a target dose of 300 mg, daily
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: sparsentan — Double-blind period: target dose of 800 mg daily; Open-label extension: target dose based on dosage from week 114 daily
  Other Names: RE-021
  Arms: sparsentan for double-blind and open-label extension
Drug: Irbesartan — target dose of 300 mg daily
  Other Names: Irbesartan Tablets USP
  Arms: Irbesartan

SUMMARY:
To determine the long-term nephroprotective potential of treatment with sparsentan as compared to an angiotensin receptor blocker in patients with primary and genetic focal segmental glomerulosclerosis (FSGS).

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind, parallel, active-control study. Approximately 300 patients aged 8 to 75 years (inclusive) will be enrolled in the study. The study will be conducted in approximately 300 study centers, globally. The investigational drug (sparsentan) is a dual-acting angiotensin receptor blocker and endothelin receptor antagonist. The active control is irbesartan. Patients who meet eligibility criteria will require washout from renin-angiotensin-aldosterone system (RAAS) blockers, if applicable prior to their first dose of study drug.

Patients will be randomly assigned in a 1:1 ratio to receive either sparsentan or active control (irbesartan).

After completing the double-blind portion of the study, patients may participate in the open-label extension for treatment with sparsentan if they meet eligibility criteria.

Primary completion date represents the anticipated completion date of the double-blind portion of the study. Study completion date represents the anticipated completion date of the open-label extension portion of the study.

ELIGIBILITY:
Key Inclusion Criteria for the Double-blind Period:

* Sites within the US and UK: The patient is male or female aged 8 to 75 years, inclusive, weighing ≥20 kg at screening
* Sites outside the US and UK: The patient is male or female aged 18 to 75 years, inclusive, weighing ≥20 kg at screening
* Biopsy-proven focal segmental glomerulosclerosis (FSGS) lesion(s) or documentation of a genetic mutation in a podocyte protein associated with FSGS.
* Urine protein/creatinine (UP/C) ≥1.5 g/g (170 mg/mmol) at screening
* eGFR ≥30 mL/min/1.73 m2 at screening.
* Women of childbearing potential must agree to the use of one highly reliable method of contraception from 7 days prior to the first dose of study medication until 90 days after the last dose of study medication, plus one additional barrier method during sexual activity

Key Exclusion Criteria for the Double-blind Period:

* FSGS secondary to another condition
* Positive serological tests of another primary or secondary glomerular disease not consistent with a diagnosis of primary or genetic FSGS
* History of type 1 diabetes mellitus, uncontrolled type 2 diabetes mellitus, or nonfasting blood glucose >180 mg/dL (10.0 mmol/L)
* Treated with rituximab, cyclophosphamide, or abatacept within ≤3 months prior to screening; if taking other chronic immunosuppressive medications, the dosage must be stable prior to screening
* Documented history of heart failure, coronary artery disease, or cerebrovascular disease
* Significant liver disease
* Positive at screening for the human immunodeficiency virus or markers indicating acute or chronic hepatitis B virus infection or hepatitis C infection
* History of malignancy other than adequately treated basal cell or squamous cell skin cancer or cervical carcinoma within the past 2 years
* Screening hematocrit value <27% (0.27 L/L) or hemoglobin value <9 g/dL (90 g/L)
* Screening potassium value of >5.5 mEq/L (5.5 mmol/L)
* Extreme obesity (ie, ≥18 years of age with a body mass index (BMI) >40, or is <18 years of age with a BMI in the 99th percentile plus 5 units at screening, in whom there is a causal relationship between obesity and the development of FSGS
* History of alcohol or illicit drug use disorder
* History of serious side effect or allergic response to any angiotensin II antagonist or endothelin receptor antagonist
* Female patient is pregnant, plans to become pregnant during the course of the study, or is breastfeeding.

Key Inclusion Criteria for the Open-label Extension Based on assessments at the Week 108 visit:

* Complete participation in the double-blind period, including the Week 112 visit.
* Patient received blinded study medication through the duration of the double-blind period (ie, did not permanently discontinue study medication)

Key Exclusion Criteria for the Open-label Extension Based on Assessments at Week 108 and 112 visits:

* Progression to end-stage renal disease requiring replacement therapy
* The patient developed criteria for discontinuation between Week 108 and Week 112
* The patient was unable to initiate, or developed contraindications to, treatment with RAAS inhibitors between Week 108 and Week 112
* eGFR ≤20 mL/min/1.73 m2 at Week 108

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Radko Komers, MD, PhD, Study Director — Travere Therapeutics, Inc.
Locations (192):
- United States (75):
  - Travere Investigational Site, Mesa, Arizona
  - Travere Investigational Site, Phoenix, Arizona
  - Travere Investigational Site, Los Angeles, California
  - Travere Investigational Site, Northridge, California
  - Travere Investigational Site, Palo Alto, California
  - Travere Investigational Site, San Diego, California
  - Travere Investigational Site, San Dimas, California
  - Travere Investigational Site, San Francisco, California
  - Travere Investigational Site, Torrance, California
  - Travere Investigational Site, Victorville, California
  - Travere Investigational Site, Denver, Colorado
  - Travere Investigational Site, Middlebury, Connecticut
  - Travere Investigational Site, Wilmington, Delaware
  - Travere Investigational Site, Washington D.C., District of Columbia
  - Travere Investigational Site, Coral Springs, Florida
  - Travere Investigational Site, Fort Lauderdale, Florida
  - Travere Investigational Site, Gainesville, Florida
  - Travere Investigational Site, Miami, Florida
  - Travere Investigational Site, Ocala, Florida
  - Travere Investigational Site, Orlando, Florida
  - Travere Investigational Site, Port Charlotte, Florida
  - Travere Investigational Site, Temple Terrace, Florida
  - Travere Investigational Site, Winter Park, Florida
  - Travere Investigational Site, Lawrenceville, Georgia
  - Travere Investigational Site, Nampa, Idaho
  - Travere Investigational Site, Chicago, Illinois
  - Travere Investigational Site, Hinsdale, Illinois
  - Travere Investigational Site, Kansas City, Kansas
  - Travere Investigational Site, Wichita, Kansas
  - Travere Investigational Site, Louisville, Kentucky
  - Travere Investigational Site, Monroe, Louisiana
  - Travere Investigational Site, New Orleans, Louisiana
  - Travere Investigational Site, Shreveport, Louisiana
  - Travere Investigational Site, Boston, Massachusetts
  - Travere Investigational Site, Springfield, Massachusetts
  - Travere Investigational Site, Ann Arbor, Michigan
  - Travere Investigational Site, Detroit, Michigan
  - Travere Investigational Site, Minneapolis, Minnesota
  - Travere Investigational Site, Rochester, Minnesota
  - Travere Investigational Site, Kansas City, Missouri
  - Travere Investigational Site, Las Vegas, Nevada
  - Travere Investigational Site, Reno, Nevada
  - Travere Investigational Site, Hackensack, New Jersey
  - Travere Investigational Site, Fresh Meadows, New York
  - Travere Investigational Site, New Hyde Park, New York
  - Travere Investigational Site, New York, New York
  - Travere Investigational Site, The Bronx, New York
  - Travere Investigational Site, Chapel Hill, North Carolina
  - Travere Investigational Site, Durham, North Carolina
  - Travere Investigational Site, Raleigh, North Carolina
  - Travere Investigational Site, Winston-Salem, North Carolina
  - Travere Investigational Site, Cleveland, Ohio
  - Travere Investigational Site, Columbus, Ohio
  - Travere Investigational Site, Oklahoma City, Oklahoma
  - Travere Investigational Site, Roseburg, Oregon
  - Travere Investigational Site, Bethlehem, Pennsylvania
  - Travere Investigational Site, Camp Hill, Pennsylvania
  - Travere Investigational Site, Philadelphia, Pennsylvania
  - Travere Investigational Site, Pittsburgh, Pennsylvania
  - Travere Investigational Site, Upland, Pennsylvania
  - Travere Investigational Site, Columbia, South Carolina
  - Travere Investigational Site, Corpus Christi, Texas
  - Travere Investigational Site, Dallas, Texas
  - Travere Investigational Site, El Paso, Texas
  - Travere Investigational Site, Fort Worth, Texas
  - Travere Investigational Site, Houston, Texas
  - Travere Investigational Site, Lewisville, Texas
  - Travere Investigational Site, Sherman, Texas
  - Travere Investigational Site, Salt Lake City, Utah
  - Travere Investigational Site, St. George, Utah
  - Travere Investigational Site, Hampton, Virginia
  - Travere Investigational Site, Spokane, Washington
  - Travere Investigational Site, Morgantown, West Virginia
  - Travere Investigational Site, Marshfield, Wisconsin
  - Travere Investigational Site, Wauwatosa, Wisconsin
- Argentina (3):
  - Travere Investigational Site, Buenos Aires
  - Travere Investigational Site, Córdoba
  - Travere Investigational Site, Santa Fe
- Australia (9):
  - Travere Investigational Site, Concord, New South Wales
  - Travere Investigational Site, New Lambton Heights, New South Wales
  - Travere Investigational Site, Saint Leonards, New South Wales
  - Travere Investigational Site, Wollongong, New South Wales
  - Travere Investigational Site, Birtinya, Queensland
  - Travere Investigational Site, Woolloongabba, Queensland
  - Travere Investigational Site, Adelaide, South Australia
  - Travere Investigational Site, Parkville, Victoria
  - Travere Investigational Site, Nedlands, Western Australia
- Belgium (3):
  - Travere Investigational Site, Leuven
  - Travere Investigational Site, Liège
  - Travere Investigational Site, Roeselare
- Brazil (7):
  - Travere Investigational Site, Botucatu
  - Travere Investigational Site, Itaquera
  - Travere Investigational Site, Passo Fundo
  - Travere Investigational Site, Porto Alegre
  - Travere Investigational Site, Recife
  - Travere Investigational Site, Rio de Janeiro
  - Travere Investigational Site, São Paulo
- Canada (3):
  - Travere Investigational Site, Edmonton, Alberta
  - Travere Investigational Site, London, Ontario
  - Travere Investigational Site, Greenfield Park, Quebec
- Travere Investigational Site, Zagreb, Croatia
- Czechia (2):
  - Travere Investigational Site, Prague, Prague
  - Travere Investigational Site, Nový Jičín
- Denmark (2):
  - Travere Investigational Site, Aarhus, Central Jutland
  - Travere Investigational Site, Kolding, Southern Denmark
- Estonia (2):
  - Travere Investigational Site, Tallinn
  - Travere Investigational Site, Tartu
- France (10):
  - Travere Investigational Site, Bordeaux
  - Travere Investigational Site, Clermont-Ferrand
  - Travere Investigational Site, Créteil
  - Travere Investigational Site, Grenoble
  - Travere Investigational Site, Marseille
  - Travere Investigational Site, Nice
  - Travere Investigational Site, Paris
  - Travere Investigational Site, Saint-Priest-en-Jarez
  - Travere Investigational Site, Toulouse
  - Travere Investigational Site, Valenciennes
- Germany (6):
  - Travere Investigational Site, Düsseldorf, Westfalen
  - Travere Investigational Site, Aachen
  - Travere Investigational Site, Berlin
  - Travere Investigational Site, Hanover
  - Travere Investigational Site, Stuttgart
  - Travere Investigational Site, Villingen-Schwenningen
- Hong Kong (2):
  - Travere Investigational Site, Hong Kong
  - Travere Investigational Site, Lai Chi Kok
- Italy (12):
  - Travere Investigational Site, Bari
  - Travere Investigational Site, Bergamo
  - Travere Investigational Site, Bologna
  - Travere Investigational Site, Florence
  - Travere Investigational Site, Genova
  - Travere Investigational Site, Germaneto
  - Travere Investigational Site, Lecco
  - Travere Investigational Site, Milan
  - Travere Investigational Site, Monza
  - Travere Investigational Site, Pavia
  - Travere Investigational Site, Roma
  - Travere Investigational Site, Verona
- New Zealand (2):
  - Travere Investigational Site, Auckland
  - Travere Investigational Site, Hamilton
- Poland (5):
  - Travere Investigational Site, Lodz
  - Travere Investigational Site, Olsztyn
  - Travere Investigational Site, Piotrkow Trybunalski
  - Travere Investigational Site, Warsaw
  - Travere Investigational Site, Wroclaw
- Portugal (7):
  - Travere Investigational Site, Amadora
  - Travere Investigational Site, Carnaxide
  - Travere Investigational Site, Lisbon
  - Travere Investigational Site, Loures
  - Travere Investigational Site, Porto
  - Travere Investigational Site, Setúbal
  - Travere Investigational Site, Vila Nova de Gaia
- South Korea (4):
  - Travere Investigational Site, Busan
  - Travere Investigational Site, Daejeon
  - Travere Investigational Site, Gyeonggi-do
  - Travere Investigational Site, Seoul
- Spain (14):
  - Travere Investigational Site, Palma de Mallorca, Balearic Islands
  - Travere Investigational Site, Lugo, Burela
  - Travere Investigational Site, Sagunto, Valencia
  - Travere Investigational Site, Badalona
  - Travere Investigational Site, Barcelona
  - Travere Investigational Site, Ciudad Real
  - Travere Investigational Site, Córdoba
  - Travere Investigational Site, Madrid
  - Travere Investigational Site, Majadahonda
  - Travere Investigational Site, Málaga
  - Travere Investigational Site, Santiago de Compostela
  - Travere Investigational Site, Seville
  - Travere Investigational Site, Valencia
  - Travere Investigational Site, Zaragoza
- Sweden (2):
  - Travere Investigational Site, Solna
  - Travere Investigational Site, Uppsala
- Taiwan (7):
  - Travere Investigational Site, Hualien City
  - Travere Investigational Site, Kaohsiung City
  - Travere Investigational Site, New Taipei City
  - Travere Investigational Site, Taichung
  - Travere Investigational Site, Tainan
  - Travere Investigational Site, Taipei
  - Travere Investigational Site, Taoyuan District
- United Kingdom (14):
  - Travere Investigational Site, Carshalton, London
  - Travere Investigational Site, Whitechapel, London
  - Travere Investigational Site, Fulwood, Preston
  - Travere Investigational Site, Brighton
  - Travere Investigational Site, Cambridge
  - Travere Investigational Site, Cardiff
  - Travere Investigational Site, Leicester
  - Travere Investigational Site, London
  - Travere Investigational Site, Manchester
  - Travere Investigational Site, Newcastle
  - Travere Investigational Site, Reading
  - Travere Investigational Site, Salford
  - Travere Investigational Site, Swansea
  - Travere Investigational Site, York

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.

REFERENCES:
- [Derived] Yee J, Gong W, Inrig J, Rheault MN, Gruber AJ, Bedard PW, Komers R, Trachtman H. Antiproteinuric Effect of Sparsentan in Patients with Genetic-Associated FSGS Enrolled in the DUPLEX Trial. Clin J Am Soc Nephrol. 2025 Dec 23. doi: 10.2215/CJN.0000000948. Online ahead of print. No abstract available. PMID 41433094
- [Derived] Rheault MN. Treatment Approaches for Alport Syndrome. J Am Soc Nephrol. 2025 Sep 12;37(1):172-9. doi: 10.1681/ASN.0000000897. Online ahead of print. PMID 40938675
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980
- [Derived] Rheault MN, Alpers CE, Barratt J, Bieler S, Canetta P, Chae DW, Coppock G, Diva U, Gesualdo L, Heerspink HJL, Inrig JK, Kirsztajn GM, Kohan D, Komers R, Kooienga LA, Lieberman K, Mercer A, Noronha IL, Perkovic V, Radhakrishnan J, Rote W, Rovin B, Tesar V, Trimarchi H, Tumlin J, Wong MG, Trachtman H; DUPRO Steering Committee and DUPLEX Investigators. Sparsentan versus Irbesartan in Focal Segmental Glomerulosclerosis. N Engl J Med. 2023 Dec 28;389(26):2436-2445. doi: 10.1056/NEJMoa2308550. Epub 2023 Nov 3. PMID 37921461
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732
- See also: Corporate Website — http://travere.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The DUPLEX study is a 112-week, Phase 3, randomized, multicenter, double-blind (DB), parallel, active-control study that evaluated the safety, tolerability, and long-term nephroprotective potential of treatment with sparsentan as compared to irbesartan in participants with focal segmental glomerulosclerosis (FSGS).
Pre-assignment Details: The study included participants 8 to 75 years of age from the United States (US) and United Kingdom (UK), and participants 18 to 75 years of age from countries other than the US and UK. The results presented are based on the primary analysis.
Groups:
- Sparsentan: Participants were randomized to receive initial dose of sparsentan as 400 milligrams (mg) over-encapsulated (blinded) with size 00 capsules orally once daily. A dose adjustment was made for participants whose body weight was ≤50 kilograms (kg) at screening; these participants received one-half of the specified dose of sparsentan. The dose was then titrated to achieve the maximum daily target dose of 800 mg.
- Irbesartan: Participants were randomized to receive active control doses of irbesartan 150 mg over-encapsulated (blinded) with size 00 capsules orally once daily. A dose adjustment was made for participants whose body weight was ≤50 kg at screening; these participants received one-half of the specified dose of irbesartan. The dose was then titrated to achieve the maximum daily target dose of 300 mg.
Period: Overall Study
Arm/Group | Sparsentan | Irbesartan
Started | 184 | 187
Completed (The participant flow presented is based on the primary analysis (double-blind period of the study).) | 168 | 171
Not Completed | 16 | 16
Not completed — Death | 4 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 7 | 11

BASELINE CHARACTERISTICS:
Population: Full Analysis Set comprised of all participants who were randomized and received at least one dose of double-blind study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sparsentan | Irbesartan | Total
Number analyzed (Participants) | 184 | 187 | 371
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.7 (16.53) | 41.5 (17.25) | 41.6 (16.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 88 | 171
  Male | 101 | 99 | 200
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 44 | 78
  Not Hispanic or Latino | 147 | 135 | 282
  Unknown or Not Reported | 3 | 8 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 23 | 27 | 50
  Black or African American | 16 | 9 | 25
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  White | 134 | 135 | 269
  Other | 5 | 12 | 17
  Multiple | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Slope of Estimated Glomerular Filtration Rate (eGFR)
Description: The total eGFR slope over 2 years, defined as the slope of eGFR following initiation of randomized treatment (ie, Day 1 to Week 108). Estimates are calculated from a mixed-effects model with treatment, Baseline eGFR, analysis visit, treatment-by-analysis visit, randomization stratification factors as fixed effects, and intercept and slope for each participant as a random effect.
Time Frame: From Day 1 to Week 108
Population: Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters/minute/1.73square meter/year
Arm/Group | Sparsentan | Irbesartan
Number analyzed (Participants) | 184 | 187
milliliters/minute/1.73square meter/year | -5.4 [-6.89 to -3.93] | -5.7 [-7.20 to -4.29]
Statistical Analysis 1: Comparison: Sparsentan vs Irbesartan; Test type: Other; p = 0.7491, Mixed Models Analysis; Slope difference = 0.3, 95% CI 2-sided [-1.74 to 2.41], Standard Error of Mean 1.05

2. Primary Outcome: Percentage of Participants Achieving FSGS Partial Remission Endpoint (FPRE)
Description: Percentage of participants achieving FPRE, defined as urine protein-to-creatinine ratio (UP/C) ≤1.5 grams/gram (g/g) (170 milligrams per millimoles [mg/mmol]) and a >40% reduction from Baseline was analyzed using a generalized linear model to model probability of achieving FPRE. Missing responses were imputed prior to analysis using multiple imputation. A generalized linear model with appropriate link function was implemented with Baseline log (UP/C), treatment, analysis visit, treatment by analysis visit interaction, and randomization strata as fixed effects. For estimates of probability of achieving FPRE, risk difference, and odds ratio, binomial distribution with logit link was used. For relative risk, Poisson distribution with log link was used. Using Rubin's approach, estimated treatment effects are combined across all imputations to obtain overall estimates for probabilities.
Time Frame: Week 36
Population: Full Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Sparsentan | Irbesartan
Number analyzed (Participants) | 184 | 187
Percentage of participants | 42.0 | 26.0
Statistical Analysis 1: Comparison: Sparsentan vs Irbesartan; Test type: Other; p = 0.0094, Mixed Models Analysis; Risk Difference (RD) = 16.00, 95% CI 2-sided [3.96 to 28.04]

3. Secondary Outcome: Slope of eGFR Following the Initial Acute Effect of Randomized Treatment
Description: The chronic eGFR slope over 2 years, defined as the slope of eGFR following the initial acute effect of randomized treatment (ie, Week 6 to Week 108). Estimates were calculated from a mixed-effects model with linear spline (ie, change point at Week 6), which included treatment, Baseline eGFR, time from Baseline (TFB) (weeks), time from change point (TFCP) (weeks), treatment-by-TFB and treatment-by-TFCP interactions, and randomization stratification factors as fixed effects, intercept and slopes as random effects. The slope difference was tested by the null hypothesis that the sum of the treatment-by-TFB and treatment-by-TFCP interactions = 0.
Time Frame: From Week 6 to Week 108
Population: Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters/minute/1.73square meter/year
Arm/Group | Sparsentan | Irbesartan
Number analyzed (Participants) | 184 | 187
milliliters/minute/1.73square meter/year | -4.8 [-6.34 to -3.27] | -5.7 [-7.20 to -4.18]
Statistical Analysis 1: Comparison: Sparsentan vs Irbesartan; Test type: Other; p = 0.4203, Mixed Models Analysis; Slope difference = 0.9, 95% CI 2-sided [-1.27 to 3.04], Standard Error of Mean 1.09

4. Secondary Outcome: Change From Baseline in eGFR to 4 Weeks Post-cessation of Randomized Treatment
Description: The change from Baseline to 4 weeks post-cessation of randomized treatment (Week 112) was analyzed via an analysis of covariance (ANCOVA) model on the natural log(eGFR) with treatment, Baseline eGFR, and randomization strata as fixed effects. Only participants who completed the 108-week treatment period were included. Estimated LS Mean and 95% CI are converted to percentages as follows: [exponential (LS mean change from baseline in natural log(eGFR)) minus 1] multiplied by 100. Baseline (Day 1) was defined as the last non-missing assessment prior to and including the first administration of study medication in the study including unscheduled assessments. Percent change from Baseline was calculated as "[(Post Baseline minus Baseline value)/ Baseline value] multiplied by 100.
Time Frame: Baseline (Day 1) to Week 112
Population: Full Analysis Set (Patients who Completed Blinded Treatment). Only those participants with data available at specified time points have been presented.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: milliliters/minute/1.73square meter
Arm/Group | Sparsentan | Irbesartan
Number analyzed (Participants) | 129 | 136
milliliters/minute/1.73square meter | -10.4 [-12.60 to -8.13] | -12.1 [-14.36 to -9.91]
Statistical Analysis 1: Comparison: Sparsentan vs Irbesartan; Test type: Other; p = 0.2708, ANCOVA; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-1.39 to 4.93]

ADVERSE EVENTS:
Time Frame: Up to Week 112
Description: Safety Analysis Set comprised of all participants who were randomized to receive at least 1 dose of double-blind study medication. The results presented are based on the primary analysis.
Groups:
- Sparsentan: Participants in this arm were randomized to receive initial dose of Sparsentan as 400 milligrams (mg) over-encapsulated (blinded) with size 00 capsules orally once daily. A dose adjustment was made for participants whose body weight was ≤50 kilograms (kg) at screening; these participants received one-half of the specified dose of Sparsentan. The dose was then titrated to achieve the maximum daily target dose of 800 mg.
Arm/Group | Sparsentan | Irbesartan
All-Cause Mortality (participants affected / at risk) | 4/184 | 3/187
Serious Adverse Events (participants affected / at risk) | 68/184 | 82/187
Other Adverse Events (participants affected / at risk) | 172/184 | 174/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sparsentan (N=184) | Irbesartan (N=187)
COVID-19 (Infections and infestations) | 22 | 39
Pneumonia (Infections and infestations) | 3 | 2
COVID-19 pneumonia (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 3
Appendicitis (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Rhinovirus infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Enterovirus infection (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1
Mycoplasma infection (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 11 | 13
Nephrotic syndrome (Renal and urinary disorders) | 5 | 3
Acute kidney injury (Renal and urinary disorders) | 3 | 8
Renal impairment (Renal and urinary disorders) | 3 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 2 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal haematoma (Renal and urinary disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 3 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 5
Generalised oedema (General disorders) | 1 | 2
Face oedema (General disorders) | 0 | 2
Peripheral swelling (General disorders) | 0 | 2
Pyrexia (General disorders) | 2 | 0
Inflammation (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 0
Swelling face (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Neonatal intestinal perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Inflammatory marker increased (Investigations) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 0 | 1
Blindness transient (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Normal labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sparsentan (N=184) | Irbesartan (N=187)
COVID-19 (Infections and infestations) | 41 | 50
Upper respiratory tract infection (Infections and infestations) | 10 | 16
Urinary tract infection (Infections and infestations) | 9 | 17
Nasopharyngitis (Infections and infestations) | 11 | 9
Influenza (Infections and infestations) | 6 | 12
Gastroenteritis (Infections and infestations) | 6 | 10
Sinusitis (Infections and infestations) | 9 | 3
Diarrhoea (Gastrointestinal disorders) | 25 | 27
Nausea (Gastrointestinal disorders) | 10 | 18
Vomiting (Gastrointestinal disorders) | 13 | 8
Abdominal pain (Gastrointestinal disorders) | 8 | 10
Abdominal pain upper (Gastrointestinal disorders) | 7 | 11
Dyspepsia (Gastrointestinal disorders) | 8 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 31 | 20
Gout (Metabolism and nutrition disorders) | 9 | 7
Oedema peripheral (General disorders) | 36 | 41
Fatigue (General disorders) | 16 | 11
Pyrexia (General disorders) | 13 | 9
Blood creatine phosphokinase increased (Investigations) | 19 | 8
Blood creatinine increased (Investigations) | 12 | 14
Glomerular filtration rate decreased (Investigations) | 12 | 11
Lipase increased (Investigations) | 8 | 11
Alanine aminotransferase increased (Investigations) | 10 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 4
Hypotension (Vascular disorders) | 33 | 21
Hypertension (Vascular disorders) | 20 | 24
Chronic kidney disease (Renal and urinary disorders) | 13 | 22
Acute kidney injury (Renal and urinary disorders) | 8 | 13
Nephrotic syndrome (Renal and urinary disorders) | 10 | 8
Proteinuria (Renal and urinary disorders) | 7 | 11
Renal impairment (Renal and urinary disorders) | 11 | 5
Dizziness (Nervous system disorders) | 23 | 21
Headache (Nervous system disorders) | 20 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Vaccination complication (Injury, poisoning and procedural complications) | 12 | 11
Anaemia (Blood and lymphatic system disorders) | 24 | 10
Anxiety (Psychiatric disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT03493685/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT03493685/SAP_001.pdf